CLINICAL TRIAL: NCT02572700
Title: Pain Mechanisms and Ultrasonographic Inflammatory Changes as Prognostic Factors in Patients With Psoriatic Arthritis: a Prospective, Exploratory Cohort Study
Brief Title: Pain Mechanisms and Ultrasonographic Disease Activity in Psoriatic Arthritis
Acronym: PIPA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Frederiksberg University Hospital (Other)
Responsible Party: Principal Investigator, Henning Bliddal, Professor, University Hospital Bispebjerg and Frederiksberg
Other Study IDs: H-15009080
Record Dates: First submitted 2015-10-02; First posted 2015-10-09 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Psoriatic Arthritis; Psoriasis; Healthy Controls
Keywords: Psoriatic arthritis; Psoriasis; DMARD; Pain; Comorbidities; Ultrasound; Immunology; Patient-reported outcomes
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis; Pain | interventions — Restraint, Physical; Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood are processed for storage in a project biobank including plasma, serum and blood leucocytes for assessment of immune characteristics and mechanisms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with psoriatic arthritis: PsA patients initiating anti-rheumatic treatment in routine care will be included as one group in the observational study. Analyses will be carried out for the overall study population as well as for subgroups (e.g., stratified according to treatment intervention) in an exploratory manner.
  Interventions: Other: Clinical examination, blood sampling, ultrasonic assessment, and questionnaires
- Patients with skin psoriasis without arthrits: 20 patients with skin psoriasis without arthrits will be included as one group at baseline only. Baseline characteristics including status of pain, fatigue, work, comorbidity and lifestyle factors will be recorded.
  Interventions: Other: Clinical examination, blood sampling, ultrasonic assessment, and questionnaires
- Healthy controls: 20 healthy controls will be included as one group at baseline only. Baseline characteristics including status of pain, fatigue, work, comorbidity and lifestyle factors will be recorded.
  Interventions: Other: Clinical examination, blood sampling, ultrasonic assessment, and questionnaires

INTERVENTIONS:
Other: Clinical examination, blood sampling, ultrasonic assessment, and questionnaires — Visits include clinical examination, questionnaires (pain, comorbidity, lifestyle, work status) and ultrasonography of joints and entheses, blood samples, and only at baseline x-ray of hands and feet.

SUMMARY:
The objective of the study is to investigate pain mechanisms, comorbidity status, biomarkers, patient reported outcome measures, ultrasonographic (US) inflammatory activity and association between these features in patients with psoriatic arthritis (PsA) intensifying anti-rheumatic treatment. Furthermore, to assess the predictive value of baseline pain profile, comorbidity status, and US joint/entheses activity on treatment outcome after 4 months. Finally, we aimed to compare baseline characteristics with I) patients with skin psoriasis without arthritis and II) healthy controls.

DETAILED DESCRIPTION:
Patients with psoriatic arthritis, who initiate or switch anti-rheumatic treatment (conventional disease modifying drugs or biologic drugs) in routine care due to an active disease state, will be enrolled in the observational study.

The overall aim is to investigate pain mechanisms, comorbidities and US psoriatic changes and elucidate if these factors - independently or by interaction - influence treatment response after 4 months. Patients will have a baseline visit, a follow up visit after 4 months and yearly thereafter. Examinations will be performed at all time points (except stated otherwise) and include:

1. Assessment of pain mechanisms by clinical evaluation (swollen/tender joint ratio, tender points) and pain questionnaires (widespread pain index, PainDETECT).
2. Ultrasonography of joints and entheses by two trained assessors
3. Clinical examination of all psoriatic manifestations
4. Interview and questionnaires regarding lifestyle, comorbidity status, function, quality of life and the impact of psoriatic manifestations.
5. Blood samples for standard rheumatic monitoring and biobank
6. X-ray of hands and feet (only at baseline)
7. AMPS test (assessment of motor and process skills) will be performed and interpreted by an certified ergo therapist (only at baseline visit and at 34-months follow-up and oly for the first included 20 PsA patients)

Clinical as well as patient-reported and observer-based outcomes will be described for the overall study population and the prognostic influence of US, comorbidities, and pain mechanisms will be analysed. Subsequently, the analyses will be repeated for certain subgroups of patients (e.g., conventional drug therapy vs. biologic drug intervention) in an exploratory manner. We will compare baseline data including pain, fatigue, work, life style and comorbidity status of PsA patients before initiating new treatment with patients with skin psoriasis without arthritis and healthy controls

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PsA according to the CASPAR (The Classification of Psoriatic Arthritis) criteria
* Peripheral joint involvement.
* Minimum 18 years of age.
* Initiating or switching anti-rheumatic treatment due to active PsA.
* Signing a written informed consent.

Exclusion Criteria:

* Pregnancy
* Peripheral neuropathy
* Demyelinising disease
* Recent stroke
* Other rheumatic inflammatory diseases.
* Oral, intra-articular or intra-muscular glucocorticoids within 3 weeks prior to baseline
* Treatment with centrally acting analgesics (opioids, anti-depressants, anticonvulsants) within 1 week prior to baseline
* Treatment with mild analgesics (non-steroidal anti-inflammatory drugs, acetylsalicylic acid, acetaminophen) within 24 hours prior to baseline

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: > 18 years of age with PsA according to the CASPAR criteria who initiate or switch anti-rheumatic treatment (biologics and/or conventional synthetic DMARDs) due to active PsA in routine care.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
American college of rheumatology 20%, | 4 months from baseline
  Composite measures of improvement in disease state (20% improvement)

SECONDARY OUTCOMES:
Disease Activity Index in Psoriatic Arthritis (DAPSA) | 4 months from baseline
  A composite measure of disease activity
Minimal Disease Activity (MDA) | 4 months from baseline
  A composite measure of disease activity

OTHER OUTCOMES:
Change in swollen joint count (SJC) | 4 months from baseline
Change in tender joint count (TJC) | 4 months from baseline
Change in Spondyloarthritis Research Consortium of Canada enthesitis score (SPARCC) | 4 months from baseline
Change in The Psoriatic Arthritis Impact of Disease-score (PsAID) | 4 months from baseline
Change in Dermatology Life Quality Index (DLQI) | 4 months from baseline
Change in Assessment of Motor and Process Skills (AMPS test) | 4 months from baseline
Transition Questionnaire score (Trans-Q) | 4 months from baseline
  Patient's judgement of overall improvement during treatment
Change in PainDETECTquestionnaire score (PDQ) | 4 months from baseline
Change in Health Assessment Questionnaire disability index (HAQ) | 4 months from baseline
Change in Visual Analogue Scale (VAS) (0-100 mm) of fatigue | 4 months from baseline
Change in Visual Analogue Scale (VAS) (0-100 mm) of pain | 4 months from baseline
Change in Visual Analogue Scale (VAS) (0-100 mm) of global disease impact | 4 months from baseline
Change in score of Medical Outcomes Study Questionnaire (SF-36) for mental and physical health | 4 months from baseline
Change in psoriasis area severity index (PASI) | 4 months from baseline
Change in ultrasonography joint scores (grey scale and doppler) | 4 months from baseline
Change in ultrasonography entheses scores (grey scale and doppler) | 4 months from baseline
Change in total cholesterol (mmol/L) | 4 months from baseline
Change in body weight (kg) | 4 months from baseline
Change in c-reactive protein (mg/L) | 4 months from baseline
Change in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | 4 months from baseline
Change in Bath Ankylosing Spondylitis Functional Index (BASFI) | 4 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Lars Erik Kristensen, MD, Ph.D, Principal Investigator — The Parker Institute, Frederiksberg and Bispebjerg Hospital, Frederiksberg, Denmark
Locations (1):
- The Parker Institute, Frederiksberg and Bispebjerg Hospital, Frederiksberg, Copenhagen, Denmark

REFERENCES:
- [Derived] Skougaard M, Stisen ZR, Jorgensen TS, Egeberg A, Hansen RL, Perez-Chada LM, Mogensen M, Merola JF, Gerwien JG, Kristensen LE. Increased prevalence of sleep disturbance in psoriatic arthritis is associated with inflammatory and non-inflammatory measures. Scand J Rheumatol. 2023 May;52(3):259-267. doi: 10.1080/03009742.2022.2044116. Epub 2022 Mar 18. PMID 35302402
- [Derived] Skougaard M, Jorgensen TS, Jensen MJ, Ballegaard C, Guldberg-Moller J, Egeberg A, Christensen R, Benzin P, Stisen ZR, Merola JF, Coates LC, Strand V, Mease P, Kristensen LE. Change in psoriatic arthritis outcome measures impacts SF-36 physical and mental component scores differently: an observational cohort study. Rheumatol Adv Pract. 2021 Nov 2;5(3):rkab076. doi: 10.1093/rap/rkab076. eCollection 2021. PMID 34778701
- [Derived] Ballegaard C, Skougaard M, Guldberg-Moller J, Nissen CV, Amris K, Jorgensen TS, Dreyer L, Kristensen LE. Comorbidities, pain and fatigue in psoriatic arthritis, psoriasis and healthy controls: a clinical cohort study. Rheumatology (Oxford). 2021 Jul 1;60(7):3289-3300. doi: 10.1093/rheumatology/keaa780. PMID 33325531
- [Derived] Hojgaard P, Ellegaard K, Nielsen SM, Christensen R, Guldberg-Moller J, Ballegaard C, Dreyer L, Mease P, de Wit M, Skov L, Glintborg B, Bliddal H, Bartels EM, Amris K, Kristensen LE. Pain Mechanisms and Ultrasonic Inflammatory Activity as Prognostic Factors in Patients With Psoriatic Arthritis: A Prospective Cohort Study. Arthritis Care Res (Hoboken). 2019 Jun;71(6):798-810. doi: 10.1002/acr.23693. Epub 2019 May 2. PMID 29975012
- [Derived] Hojgaard P, Christensen R, Dreyer L, Mease P, de Wit M, Skov L, Glintborg B, Christensen AW, Ballegaard C, Bliddal H, Bukhave K, Bartels EM, Amris K, Ellegaard K, Kristensen LE. Pain mechanisms and ultrasonic inflammatory activity as prognostic factors in patients with psoriatic arthritis: protocol for a prospective, exploratory cohort study. BMJ Open. 2016 Apr 15;6(4):e010650. doi: 10.1136/bmjopen-2015-010650. PMID 27084281